CLINICAL TRIAL: NCT04471987
Title: A Phase I Study to Evaluate Safety and Early Signs of Efficacy of the Human Monoclonal Antibody-cytokine Fusion Protein IL12-L19L19.
Brief Title: Safety and Early Signs of Efficacy of IL12-L19L19.
Acronym: DODEKA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PH- IL12L19L19-01/19; 2024-510841-32-00 (EU CTIS Number)
Record Dates: First submitted 2020-07-07; First posted 2020-07-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, non-randomized, multiple ascending dose, phase I dose escalation trial in patients with advanced solid carcinomas after previous immune-checkpoint blockade therapy conducted in sequential cohorts of patients followed by a dose expansion part.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The study will take place in two stages:
  1. In the dose escalation part, participants will be enrolled in cohorts and will be treated with different doses of IL12-L19L19 in order to identify a RD to be further explored in the subsequent dose expansion part. In the dose escalation part, patients will be treated in cohorts of 1 to 6 patients with escalating doses of IL12-L19L19 until the MAD is reached.
  2. Following successful identification of the RD, the study will proceed with a dose expansion part and 20 patients will be treated at the RD dose level.
  Interventions: Drug: IL12-L19L19

INTERVENTIONS:
Drug: IL12-L19L19 — Part I - The dose escalation is designed with an initial accelerated phase followed by a standard 3+3 design. Cohorts contain one patient until first instance of moderate toxicity or a DLT in the DLT observation period (28 days). With the second occurrence of moderate toxicity or occurrence of a DLT the accelerated phase will be terminated and the dose escalation will continue with a 3+3 dose escalation. Initiation of the study treatment for an individual subject will occur not less than 7 days after initiation of the study treatment for the previous patient. Not more than 2 patients are to be treated simultaneously within their DLT observation period (i.e., Day 1 to Day 28).
  Part II - Dose expansion: Once the dose escalation is completed, additional 20 patients will be enrolled at the RD to better understand the safety profile and to explore early signs of efficacy in different disease indications.
  Other Names: Dodekin
Drug: IL12-L19L19 — Patients initially receive 8 consecutive administrations of IL12-L19L19 every week. At the end of this eight weeks treatment window, a tumor assessment is performed and those patients who achieve a clinical benefit (SD, PR, CR) may continue treatment with IL12-L19L19 as a biweekly maintenance therapy until disease progression, unacceptable toxicity, withdrawal of consent, at the discretion of the investigator or up to 1 year from study treatment start.
  Other Names: Dodekin

SUMMARY:
The purpose of this study is to describe the safety, tolerability and early signs of efficacy of the antibody-cytokine fusion protein IL12-L19L19 in patients with advanced or metastatic solid carcinomas, after previous immune checkpoint blockade therapy.

The primary objective of the study is to evaluate the safety of IL12-L19L19 and to establish MTD in order to establish a recommended dose (RD).

The secondary objectives of the study are to assess early signs of efficacy, the determination of pharmacokinetic (PK) properties and the immunogenicity of IL12-L19L19.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged 18 to 80 years at the time of consent.
2. Patients must have a histological or cytological diagnosis of advanced/metastatic immunotherapy responsive solid carcinoma for which immune checkpoint blockade is approved, that has progressed on immune checkpoint-blockade therapy.
3. Patients must have received an immune checkpoint blockade therapy-based regimen as prior treatment.
4. Only patients without other therapeutic alternatives with curative or survival prolonging potential per investigator judgement are able to participate.
5. Subjects must have had clinical benefit in terms of disease control (CR/PR/SD) while on checkpoint inhibitor treatment defined as ≥ 3 month free from progression from initial imaging documenting advanced/metastatic disease followed by radiographic disease progression after checkpoint inhibitor per investigator's opinion.
6. Patients must have progressive disease or relapse at the time of screening.
7. Patients may have previously received chemotherapy, immunotherapy or radiation therapy. Such therapies must be completed at least 4 weeks prior to study drug administration. Radiotherapy within 4 weeks of the first dose of study drug, is allowed for palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass. During the expansion part, to allow evaluation of response to treatment, patients must have remaining measurable disease that has not been irradiated.
8. Eastern cooperative oncology group (ECOG) performance status ≤ 2.
9. Patient has an estimated life expectancy of at least 12 weeks.
10. At least one unidimensionally measurable lesion either by computed tomography (CT), MRI or PET/CT as defined by RECIST (v. 1.1) for solid tumors.
11. Documented negative test for HIV-HBV-HCV. For HBV serology: the determination of HBsAg, and anti-HBcAg-Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required. For HCV: HCV-RNA or HCV antibody test. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
12. All acute toxic effects (excluding alopecia and fatigue) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v. 5.0) Grade ≤ 1.
13. Full resolution of checkpoint blockade therapy-related adverse effects (including immune-related adverse effects) and no treatment for these AEs for at least 4 weeks prior to the time of enrollment. The only exception are patients with checkpoint blockade induced hypothyroidism and hypophysitis if these patients are on stable maintenance therapy with on levothyroxine or steroids (≤ 10 mg prednisone equivalent) for at least 2 months prior dosing.
14. No history of severe immune related adverse effects from prior given immune checkpoint blockade therapy (CTCAE Grade 4; CTCAE Grade 3 requiring treatment >4 weeks).
15. Female patients: negative blood pregnancy test at Screening for women of childbearing potential (WOCBP)*. WOCBP must agree to use, from the screening to six months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.
16. Male patients: male subjects able to father children must agree to use two acceptable methods of contraception throughout the study (e.g. condom with spermicidal gel). Double-barrier contraception is required.
17. Negative TB test (e.g. Mantoux or Quantiferon assay).
18. A personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study and has given consent to participate in the study.
19. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

    * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy)

Exclusion Criteria:

1. Subjects who participated in an investigational drug or device study within 4 weeks prior to study treatment start.
2. Radiotherapy within 4 weeks prior to study treatment start.
3. Active or history of autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent.
4. Patients with primary brain tumors or CNS disease (including brain metastases).
5. Patient taking herbal medications within 7 days prior to study treatment start.
6. Known history of allergy to an excipient in study medication or any other intravenously administered human proteins/peptides/antibodies.
7. Absolute neutrophil count (ANC) < 1.5 x 10^9/L, platelets < 100 x 10^9/L or haemoglobin (Hb) < 9.0 g/dl.
8. Chronically impaired renal function as indicated by creatinine clearance < 60 mL/min or serum creatinine > 1.5 ULN.
9. Inadequate liver function (ALT, AST, ALP ≥ 2.5 x ULN or total bilirubin ≥ 2.0 x ULN). At the discretion of the investigator, an increased exclusion threshold for patients with liver metastasis can be accepted as follows: ALT, AST, ALP and bilirubin ≥ 5 x ULN.
10. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol, in the opinion of the investigator.
11. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
12. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
13. Clinically significant cardiac arrhythmias or requiring permanent medication.
14. Abnormal LVEF or any other abnormalities observed during baseline ECG and echocardiogram investigations that are considered as clinically significant by the investigator. Subjects with current, or a history of QT/QTc prolongation would be excluded. In particular:

    * patients with a marked prolongation of QT/QTc interval (e.g., repeated demonstration of QTc >480 milliseconds using Fredricia's QT correction formula) are excluded;
    * patients with a history of risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of prolonged QT syndrome) are excluded;
    * patients who require the use of concomitant medications that prolong the QT/QTc interval are excluded.
15. Uncontrolled hypertension as defined by systolic blood pressure ≥ 140 mmHg and diastolic blood pressure ≥ 90 mmHg at 3 consecutive measurements performed within one week. Note: if the first blood pressure measurement is below threshold for systolic or diastolic blood pressure, it is not required to repeat the measurement.
16. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
17. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
18. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of study treatment start.
19. Pregnancy or breast-feeding.
20. Systemic chronic steroid therapy (>10 mg/day prednisone or equivalent) or any other immunosuppressive therapy within 14 days prior to study treatment start. Topical, inhaled, nasal and ophthalmic steroids are allowed.
21. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
22. Concurrent or previous malignancies (other than the indication for this trial), unless a complete remission without further recurrence was achieved at least 2 years prior to study treatment start.
23. Growth factors or immunomodulatory agents within 7 days prior to study treatment start.
24. Serious, non-healing wound, ulcer or bone fracture.
25. Deep vein thrombosis, pulmonary embolism or other acute vascular events within 6 months.
26. Requirement of concurrent use of other anti-cancer treatments or agents other than study medication.
27. Any recent live vaccination within 4 weeks prior to treatment or plan to receive vaccination during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
For Part I: DLT | From Day 1 to Day 28 of the treatment
  Occurrence of dose limiting toxicity (DLT) in dose escalation part of the study.
For Part I: MAD | From Day 1 to Day 28 of the treatment
  Definition of Maximum Administered Dose (MAD) (in dose escalation part). The MAD is defined when at least two patients within a cohort of 2-6 patients experience a DLT (i.e., ≥33% of patients with a DLT at that dose level)
For Part I: MTD and RD | From Day 1 to Day 28 of the treatment
  Defining the Maximum Tolerated Dose (MTD) and recommendation of the Recommended Dose (RD): when the DLT rate reaches 33% in a cohort, the next lower dose level will be called the MTD (so long as the DLT rate is less than 33%). Accordingly, the recommended dose (RD) for the Dose Expansion cohort will be the MTD.
Safety (AE) | Throughout study completion for each patient
  Safety of administration of IL12-L19L19, through an assessed by Common Toxicity Criteria (version 5.0, CTCAE)
Safety (SAE) | Throughout study completion for each patient
  Safety of administration of IL12-L19L19, assessed by Common Toxicity Criteria (version 5.0, CTCAE)
Safety (DILI) | Throughout study completion for each patient, a maximum of 24 weeks for each patient
  Evaluation of possible Drug Induce Liver Injury, caused by IL12-L19L19, assessed by Common Toxicity Criteria (version 5.0, CTCAE)

SECONDARY OUTCOMES:
Plasma concentration of IL12-L19L19 | 30 min prior injection in week from 1 to 8, at End-of-Treatment Visit and Follow Up 1; in week 1 and 3: 15 min after start of infusion, 60 min after start of infusion, end of infusion, 2h, 4h and 24h after end of infusion
  Evaluation of individual plasma concentration of IL12-L19L19
AUC of IL12-L19L19 | In week 1 and 3: 15 min after start of infusion, 60 min after start of infusion, end of infusion, 2 h after end of infusion, 4 h after end of infusion, 24 h after end of infusion
  Estimation of AUC of IL12-L19L19, as data permit
Tmax of IL12-L19L19 | In week 1 and 3: 15 min after start of infusion, 60 min after start of infusion, end of infusion, 2 h after end of infusion, 4 h after end of infusion, 24 h after end of infusion
  Estimation of Tmax of IL12-L19L19, as data permit
T1/2 of IL12-L19L19 | in week 1 and 3: 15 min after start of infusion, 60 min after start of infusion, end of infusion, 2 h after end of infusion, 4 h after end of infusion, 24 h after end of infusion
  Estimation of T1/2 of IL12-L19L19, as data permit
Cmax of IL12-L19L19 | in week 1 and 3: 15 min after start of infusion, 60 min after start of infusion, end of infusion, 2 h after end of infusion, 4 h after end of infusion, 24 h after end of infusion
  Estimation of Cmax of IL12-L19L19, as data permit
HAFA | At week 1, 2, 3 and 4
  Formation of human anti-fusion protein antibodies (HAFA) against IL12-L19L19
For Part II: ORR | At 8 weeks, 16 weeks, 24 weeks, 36 weeks and 48 weeks.
  Objective Response Rate (ORR, consisting of complete response (CR) + partial response (PR)), is defined as the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period. Response duration usually is measured from the time of initial response until documented tumor progression. ORR is the sum of partial responses (PR) plus complete responses (CR), based on Response Evaluation Criteria in Solid Tumors (RECIST) (v. 1.1) criteria.
For Part II: DoR | At 8 weeks, 16 weeks, 24 weeks, 36 weeks and 48 weeks.
  The duration of overall response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) untile the first date that recurrent or PD is objectively documented.
For Part II: PFS | At 8 weeks, 16 weeks, 24 weeks, 36 weeks and 48 weeks.
  Progression Free Survival (PFS) the time from enrolment to progression or death from any cause.
For Part II: OS | At 8 weeks, 16 weeks, 24 weeks, 36 weeks and 48 weeks.
  Overall Survival (OS) is defined beginning from enrolment to death from any cause

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (4):
  - Universitaetsklinik Hamburg-Eppendorf, Hamburg, Hamburg
  - Universitätsklinikum Heidelberg, Nationalen Centrum für Tumorerkrankungen (NCT), Dermatoonkologie, Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Klinik für Dermatologie, Venerologie und Allergologie, Leipzig, Leipzig
  - Universitätsklinikum Tübingen, Klinik für Innere Medizin VIII Medizinische Onkologie und Pneumologie, Tübingen
- Italy (3):
  - IEO - Istituto Europeo di Oncologia, Milan, Italy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano
- Switzerland (4):
  - Universitätsspital Basel, Basel, Basel
  - Insel Gruppe AG, Bern, Canton of Bern
  - Geneva University Hospital, Oncology Department, Geneva, Canton of Geneva
  - Oncology Institute of Southern Switzerland, Bellinzona

IPD SHARING:
Plan to Share IPD: No